CLINICAL TRIAL: NCT03700658
Title: A Randomized Cross-Over Study to Evaluate Local Tolerability Following Subcutaneous Administration of TV-46046
Brief Title: A Study to Evaluate Injection Pain and Local Tolerability Following Subcutaneous (SC) Administration of TV-46046
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TV46046-WH-10147
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Contraception
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Masking Description: The study will be partially blinded due to differences in appearance and volume of the treatments. Designated unblinded study staff will conduct randomization procedures. The staff preparing and administering injections will also be unblinded to treatment sequence but will be trained to shield the syringe prior to and at the time of injection from view of the participant and study staff assessing injection site reactions (ISRs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TV-46046 Undiluted (Experimental): Participants will receive TV-46046 undiluted (120 mg/0.3 mL of 400 mg/mL) SC injection as a test formulation in a crossover design with the other 3 SC study drug injections. The 4 study drug injections will be administered approximately 1 hour apart.
  Interventions: Drug: TV-46046
- TV-46046 Diluted (Experimental): Participants will receive TV-46046 saline-diluted (60 mg/0.3 mL of 200 mg/mL) SC injection as a test formulation in a crossover design with the other 3 SC study drug injections. The 4 study drug injections will be administered approximately 1 hour apart.
  Interventions: Drug: TV-46046
- TV-46046 Placebo (Placebo Comparator): Participants will receive TV-46046 placebo (0.3 mL) SC injection in a crossover design with the other 3 SC study drug injections. The 4 study drug injections will be administered approximately 1 hour apart.
  Interventions: Drug: TV-46046 Placebo
- Depo-subQ 104 (Active Comparator): Participants will receive Depo-subQ 104 (medroxyprogesterone acetate injectable suspension; 104 mg/0.65 mL) SC injection as a reference formulation in a crossover design with the other 3 SC study drug injections. The 4 study drug injections will be administered approximately 1 hour apart.
  Interventions: Drug: Depo-subQ 104

INTERVENTIONS:
Drug: TV-46046 — TV-46046 will be administered per dose and schedule specified in the arm.
  Arms: TV-46046 Diluted; TV-46046 Undiluted
Drug: Depo-subQ 104 — Depo-subQ 104 will be administered per dose and schedule specified in the arm.
  Other Names: Medroxyprogesterone acetate injectable suspension; Depo-subQ Provera 104®
  Arms: Depo-subQ 104
Drug: TV-46046 Placebo — TV-46046 Placebo will be administered per schedule specified in the arm.
  Arms: TV-46046 Placebo

SUMMARY:
The purpose of this study is to evaluate the local tolerability associated with the SC administration of TV-46046, and inform next steps of the TV-46046 development program.

DETAILED DESCRIPTION:
Eligible participants will be enrolled and receive 1 of each of the 4 SC study injections in each abdominal quadrant approximately 1 hour apart: 120 milligrams (mg)/0.3 milliliter (mL) of TV-46046, 60 mg/0.3 mL of 1:1 saline diluted TV-46046, 0.3 mL of TV-46046 Placebo and 104 mg/0.65 mL Depo-subQ 104 per the assigned sequence.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a low risk of pregnancy (that is, sterilized, in exclusively same-sex partnership, in menopause and/or post-menopausal, abstinent, in a monogamous relationship with vasectomized partner, using nonhormonal intrauterine device [IUD], or consistent use of condoms)
* Participant is not pregnant and does not have desire to become pregnant in the subsequent 18 months
* Participant had a normal mammogram within the last year, if 40 years or older
* Participant has no skin disorders or skin allergies

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Participant has hypertension
* Participant has ischemic heart disease or a history of ischemic heart disease
* Participant has a history of stroke
* Participant has a history of thromboembolic event(s)
* Participant has systemic lupus erythematosus
* Participant has rheumatoid arthritis and is undergoing immunosuppressive therapy
* Participant has migraine with aura
* Participant has unexplained vaginal bleeding
* Participant has diabetes
* Participant has a strong family history of breast cancer
* Participant has cervical cancer or a history of cervical cancer
* Participant has severe cirrhosis (decompensated) or liver tumors
* Participant has known significant renal disease
* Participant has a history of diagnosed clinical depression or bipolar disorder, with or without suicidal ideation, and/or history of suicide attempt
* Participant is currently using hormonal contraception
* Participant had an injection of DMPA (Depo-Provera CI or Depo-subQ 104) in the past 12 months; or combined injectable in the last 3 months
* Participant is chronically using pain medication
* Participant has a plan to move to another location in the next 18 months

  * Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 1, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Participants received TV-46046 undiluted (120 milligrams [mg]/0.3 milliliters [mL] of 400 mg/mL) and TV-46046 saline-diluted (60 mg/0.3 mL of 200 mg/mL) subcutaneous (SC) injection as a test formulation, Depo-subQ 104 (medroxyprogesterone acetate injectable suspension; 104 mg/0.65 mL) SC injection as a reference formulation, and TV-46046 placebo SC injection in a crossover design. The 4 study drug injections were administered approximately 1 hour apart.
Period: Overall Study
Arm/Group | Overall Study
Started | 27
Received at Least 1 Dose of Study Drug | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The treated analysis set included all participants who received at least 1 of the 4 study drug injections.
Groups:
- Overall Study: Participants received TV-46046 undiluted (120 mg/0.3 mL of 400 mg/mL) and TV-46046 saline-diluted (60 mg/0.3 mL of 200 mg/mL) SC injection as a test formulation, Depo-subQ 104 (medroxyprogesterone acetate injectable suspension; 104 mg/0.65 mL) SC injection as a reference formulation, and TV-46046 placebo SC injection in a crossover design. The 4 study drug injections were administered approximately 1 hour apart.
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (6.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Biracial | 26
  Race: Black or African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Injection Site Reactions (ISRs) (Excluding Injection Site Pain)
Description: ISRs were assessed by self-reports and direct observation for each injection at least twice on the day of injection. ISRs included erythema (redness), swelling, pruritus (itching), bleeding, bruising, injection site discoloration (for example, hypopigmentation), or atrophy (that is, dimple).
Time Frame: Day 0 (immediately after and 1 hour after the injection) up to Month 18
Population: The treated analysis set included all participants who received at least 1 of the 4 study drug injections excluding 3 participants who had partial injections.
Measure: Count of Participants; unit: Participants
Groups:
- TV-46046 Undiluted: Participants received TV-46046 undiluted (120 mg/0.3 mL of 400 mg/mL) subcutaneous (SC) injection as a test formulation.
- TV-46046 Diluted: Participants received TV-46046 saline-diluted (60 mg/0.3 mL of 200 mg/mL) SC injection as a test formulation.
- TV-46046 Placebo: Participants received TV-46046 placebo (0.3 mL) SC injection.
- Depo-subQ 104: Participants received Depo-subQ 104 (medroxyprogesterone acetate injectable suspension; 104 mg/0.65 mL) SC injection as a reference formulation.
Arm/Group | TV-46046 Undiluted | TV-46046 Diluted | TV-46046 Placebo | Depo-subQ 104
Number analyzed (Participants) | 25 | 27 | 27 | 26
Participants | 12 | 6 | 0 | 8

2. Secondary Outcome: Injection Site Pain Score, as Assessed by Numerical Rating Scale (NRS)
Description: Participants assessed their injection site pain using an 11-point NRS (0 = no pain at all; 10 = worst pain). Higher scores denote worse outcome.
Time Frame: Day 0 (Immediately after and 1 hour after injection)
Population: The treated analysis set included all participants who received at least 1 of the 4 study drug injections excluding 5 participants with needle blockage/manipulation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TV-46046 Undiluted: Participants received TV-46046 undiluted (120 mg/0.3 mL of 400 mg/mL) SC injection as a test formulation.
Arm/Group | TV-46046 Undiluted | TV-46046 Diluted | TV-46046 Placebo | Depo-subQ 104
Number analyzed (Participants) | 22 | 22 | 22 | 22
units on a scale
  Immediately after injection | 2.1 (1.72) | 1.9 (1.46) | 3.3 (2.15) | 1.2 (1.40)
  1 hour after injection | 0.2 (0.50) | 0.2 (0.50) | 0.6 (1.00) | 0.1 (0.29)

3. Secondary Outcome: Participant's Perception of Pain, as Assessed by an Overall Ranking of the 4 Study Injections From Least to Most Painful
Description: Each participant was asked to rank the injections according to overall pain from least (score = 1) to most (score = 4) painful. If a participant could not rank all of her injections from least to most painful or could not uniquely identify which injection was the most painful, then her responses were appropriately weighted across groups (for example, if a participant ranked all 4 treatments as equally most painful, then that participant contributed a score of 0.25 to each group when assessing the distribution of the most painful injection and in the event of a tie between 2 rankings, 0.5 was assigned to each tied ranking).
Time Frame: Day 0 (1 hour after injection)
Population: as for outcome 2
Measure: Number; unit: frequency (number of times) of ranking
Arm/Group | TV-46046 Undiluted | TV-46046 Diluted | TV-46046 Placebo | Depo-subQ 104
Number analyzed (Participants) | 22 | 22 | 22 | 22
frequency (number of times) of ranking
  Pain Rank 1 | 4 | 5 | 4 | 9
  Pain Rank 2 | 8.5 | 8.5 | 0 | 5
  Pain Rank 3 | 4.5 | 4.5 | 6 | 7
  Pain Rank 4 | 5 | 4 | 12 | 1

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were considered treatment emergent if (a) the onset occurred on or after the time of first injection or (b) an event had an onset prior to the first injection but increased in severity after administration of the injection. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Day 0 up to Month 18
Population: The treated analysis set included all participants who received at least 1 of the 4 study drug injections.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Participants | 23

ADVERSE EVENTS:
Time Frame: Day 0 up to Month 18
Description: The treated analysis set included all participants who received at least 1 of the 4 study injections. The adverse events which occurred during the follow-up are reported in a separate arm "Follow-up After Treatment".
Groups:
- Follow-up After Treatment: All Participants were followed for at least 6 months after receiving their injections. Participants with unresolved injection site reactions (ISRs) were followed monthly through the resolution of ISRs or Month 18, whichever came first.
- TV-46046 Undiluted: Participants received TV-46046 undiluted (120mg/0.3 mL of 400 mg/mL) SC injection as a test formulation.
- TV-46046 Placebo: Participants received TV-46046 placebo SC injection.
Arm/Group | Follow-up After Treatment | TV-46046 Undiluted | TV-46046 Diluted | TV-46046 Placebo | Depo-subQ 104
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 18/27 | 0/27 | 1/27 | 2/27 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follow-up After Treatment (N=27) | TV-46046 Undiluted (N=27) | TV-46046 Diluted (N=27) | TV-46046 Placebo (N=27) | Depo-subQ 104 (N=27)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follow-up After Treatment (N=27) | TV-46046 Undiluted (N=27) | TV-46046 Diluted (N=27) | TV-46046 Placebo (N=27) | Depo-subQ 104 (N=27)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acarodermatitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03700658/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03700658/SAP_001.pdf